CLINICAL TRIAL: NCT03325153
Title: Screening for Obstructive Sleep Apnea Predicts Cardiopulmonary Events in Patients Undergoing Bronchoscopy
Brief Title: Obstructive Sleep Apnea and Bronchoscopy
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jinwoo Lee, Associate professor, Seoul National University Hospital
Other Study IDs: 1612041813
Record Dates: First submitted 2017-10-25; First posted 2017-10-30 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Obstructive Sleep Apnea of Adult
Keywords: Obstructive Sleep Apnea; Bronchoscopy; STOP-Bang questionnaire; Cardiopulmonary events
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The prevalence of sleep-disordered breathing in Republic of Korea is 27% and 16% in men and women aged 40-69 years. Up to 93% of women and 82% of men with obstructive sleep apnea (OSA) remain undiagnosed. Polysomnography, the gold standard, is time consuming and costly. Patients with undiagnosed OSA may experience obstructive episodes during procedures with conscious sedation.

STOP-Bang questionnaire is the validated questionnaire to screen patients for undiagnosed OSA in the preoperative setting. It has high sensitivity (92.9%) for predicting patients with moderate to severe OSA.

Previous studies reported that STOP-Bang questionnaire predicted cardiopulmonary events during advanced endoscopic procedures such as endoscopic retrograde cholangiopancreatography (ERCP) and endoscopic ultrasound. However, there have been no studies regarding the risk for sedation-related cardiopulmonary events in patients with undiagnosed OSA undergoing bronchoscopy. Thus, we aimed to evaluate the prevalence of high-risk patients for OSA by a screening questionnaire, and to determine whether the questionnaire could predict patients who are at risk for cardiopulmonary events during bronchoscopy with conscious sedation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are18 years or order undergoing bronchoscopy with conscious sedation in the bronchoscopy center

Exclusion Criteria:

* Previous diagnosis of OSA
* American Society of Anesthesiologists Physical Status Classification System score > 3
* Baseline SpO2 < 90% or need for supplemental oxygen before the procedure
* Tracheostomy tubes
* An inability to provide informed consent
* Undergoing the procedure based on an outpatient clinic
* Undergoing BAL, EBUS-TBNA, and interventional bronchoscopy
* Allergies or sensitivities to sedative medications
* Pregnant

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary referral hospital
Sampling Method: Non-Probability Sample
Enrollment: 546 (Actual)
Dates: Start 2016-12-27 (Actual); Primary Completion 2018-09-21 (Actual); Study Completion 2018-12-27 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary events | Any time during bronchoscopy under conscious sedation (procedure)
  Hypoxemia (SpO2 < 90%) or Hypotension (SBP < 90 mm Hg or a decrease of more than 25% from the baseline)

SECONDARY OUTCOMES:
Airway maneuvers | Any time during bronchoscopy under conscious sedation (procedure)
  Chin lift or Bag-mask ventilation or Unplanned endotracheal intubation

CONTACTS AND LOCATIONS:
Overall Officials: Jinwoo Lee, MD, Principal Investigator — Seoul National University
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Cho J, Choi SM, Park YS, Lee CH, Lee SM, Yoo CG, Kim YW, Lee J. Prediction of cardiopulmonary events using the STOP-Bang questionnaire in patients undergoing bronchoscopy with moderate sedation. Sci Rep. 2020 Sep 2;10(1):14471. doi: 10.1038/s41598-020-71314-1. PMID 32879339